CLINICAL TRIAL: NCT01242592
Title: Homeopathy as an Adjuvant to Chemotherapy Improves Clinical Outcome in Relapsed Pulmonary Tuberculosis: Randomized Placebo Controlled Trial
Brief Title: Homeopathy as an Adjuvant to Chemotherapy Improves Clinical Outcome in Relapsed Pulmonary Tuberculosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NMP Medical Research Institute (Other)
Responsible Party: Dr Neha Sharma, NMP Medical Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NMP/H/01
Record Dates: First submitted 2010-11-16; First posted 2010-11-17 (Estimated); Last update posted 2010-11-17 (Estimated); Status verified 2010-11

CONDITIONS: Pulmonary Tuberculosis
MeSH Terms: conditions — Tuberculosis, Pulmonary

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Homeopathy (Experimental)
  Interventions: Drug: Anti-Tuberculosis Treatment
- Placebo (Placebo Comparator)
  Interventions: Drug: Anti-Tuberculosis Treatment

INTERVENTIONS:
Drug: Anti-Tuberculosis Treatment
  Other Names: DOT CAT II

SUMMARY:
The purpose of the study is to evaluate the effect of homeopathy as an adjuvant to Anti tuberculosis treatment on sputum conversion, hematological, clinical sign and symptoms of relapsed Pulmonary TB.

ELIGIBILITY:
Inclusion Criteria:

relapse pulmonary tuberculosis patients with acid-fast bacilli smear positive by microscopy, using ZiehlNieelsen staining as recommended by WHO, unfit for DOTS -

Exclusion Criteria:

pregnancy, clinical sign of any concomitant disease such as diabetes mellitus, acute renal failure or infectious disease including TB/HIV and HIV positive, currently or taken any alternative therapies in past 6 months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2005-02; Study Completion 2008-06

PRIMARY OUTCOMES:
Sputum conversion
  Sputum AFB status by microscopy will be recorded. Sputum conversion is defined as three consecutive sputum smears negative for AFB.

SECONDARY OUTCOMES:
Quality of Life
  Quality of life assessed using SF 36 questionnaire 20 before treatment and after follow up of 11 months. Low numeric scores reflect a perception of poor health, loss of function, and presence of pain

CONTACTS AND LOCATIONS:
Overall Officials: Neha Sharma, PhD, Principal Investigator — NMP Medical Research Institute
Locations (1):
- NMP medical Research Institute, Jaipur, Rajastha, India